CLINICAL TRIAL: NCT05440578
Title: Outcomes of First-line Olaparib Combined With Bevacizumab Maintenance Therapy in Newly Diagnosed Ovarian Cancer Patients With tBRCA Wild-type Tumors: a Real-world Study
Brief Title: First-line Olaparib Combined With Bevacizumab Maintenance Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-20-20889-01
Record Dates: First submitted 2021-12-08; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Neoplasms
Keywords: tBRCA， olaparib，bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- olaparib plus bevacizumab treatment group: olaparib plus bevacizumab maintenance therapy in clinical practice and will be conducted in patients with tBRCAwt newly diagnosed high grade epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy following the standard of care from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required) at tertiary-referral university hospitals and main cancer centers in China.
  Interventions: Drug: olaparib plus bevacizumab maintenance therapy

INTERVENTIONS:
Drug: olaparib plus bevacizumab maintenance therapy — First-line olaparib plus bevacizumab maintenance therapy initiated from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required).

SUMMARY:
Four phase III trials in ovarian cancer consistently showed that front-line poly(ADP-ribose) polymerase (PARP) inhibition can significantly improve progression-free survival. Based on these findings, current clinical guidelines recommend the olaparib plus bevacizumab combination as a maintenance therapy for ovarian cancer patients with BRCA1/2 wild-type or unknown mutation status who have a complete response (CR)/ partial response (PR) after completing bevacizumab-containing first-line therapy. However, bevacizumab is not a NATIONAL MEDICAL PRODUCTS ADMINSTRATION（ NMPA） -approved agent for ovarian cancer patients. In this setting, there is no olaparib plus bevacizumab maintenance therapy RWS data amongst 1st tBRCAwt patients in China, while this treatment regimen has been used in Chinese clinical practise by some doctors based on above-mentioned data.

DETAILED DESCRIPTION:
The main objective is to evaluate the outcome of olaparib plus bevacizumab combination maintenance therapy by proportion of patients alive and progression free at 1 year (1-yr PFSrate) We hypothesize that olaparib plus bevacizumab maintenance therapy could be beneficial for tBRCAwt high-grade serous ovarian cancer (HGSOC) patients who are treated with platinum-based first-line chemotherapy.

The secondary objectives are to evaluate the outcomes of olaparib plus bevacizumab maintenance therapy by: 1) 2-yr PFS rate; 2) median PFS; 3) median Time to First Subsequent Therapy or death (mTFST) ; 4) post-progression treatment after first progression; 5) reason for olaparib plus bevacizumab dose adjustment, dose interruptions, and dose discontinuations; 6) Reason for use of concomitant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients must be ≥18 years old at diagnosis.
* Patients with newly diagnosed, histologically confirmed, advanced (FIGO stage III-IV) ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer and received olaparib and plus bevacizumab from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required)
* Patients must have a tumor BRCA testing result which is tBRCAwt, defined as tumor BRCA wild type (patients without evidence of BRCA 1 and/or BRCA 2 deleterious or suspected deleterious mutations)
* Patients who have completed first-line platinum-based chemotherapy and were in clinical complete response (CR) or in partial response (PR)
* Patients who were still in CR or PR before receiving maintenance therapy
* Patients who received at least one dose of olaparib plus bevacizumab maintenance therapy within three months after platinum-based chemotherapy and without disease progression

Exclusion Criteria:

* Patient with multiple primary cancers as reported in EMR
* Concomitant any anti- cancer therapy (chemotherapy, immunotherapy, hormonal therapy (Hormone replacement therapy (HRT) is acceptable), radiotherapy, biological therapy or other novel agent) during olaparib plus bevacizumab maintenance therapy.
* Any previous treatment with PARP inhibitor.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases.
* Any other concerns related to decreased efficacy and safety of maintenance therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HGSOC who started first-line olaparib plus bevacizumab maintenance therapy from Aug 2018 up to Dec 2020 (the time range could be extended in order to recruit enough eligible subjects as required) will be identified from the electronic medical record system.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
1-yr PFS rate | 12 months after date of first dose
  the investigator assessed progression-free survival (PFS) at 1 year

SECONDARY OUTCOMES:
2-yr PFS rate | 24 months after date of first dose
  the investigator assessed progression-free survival (PFS) at 2 year
Median PFS | Median time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  median progression-free survival
mTFST | Median time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  median Time to First Subsequent Therapy or death
Post-progression treatment | Through study completion, an average of 1 year
  The proportion of patients receiving each treatment after first progression through study completion, an average of 1 year